CLINICAL TRIAL: NCT02724566
Title: Influence of Apelin on Insulin Sensitivity in Type 2 Diabetic Volunteers
Brief Title: Effect of Apelin on Insulin Sensitivity in Type 2 Diabetic Volunteers
Acronym: APELINS-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Société Francophone du Diabète (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 15 7783 03
Record Dates: First submitted 2016-03-18; First posted 2016-03-31 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2017-08

CONDITIONS: Diabetes
Keywords: Type 2 diabetic volunteers
MeSH Terms: conditions — Diabetes Mellitus | interventions — Apelin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apelin then Placebo (Other): First clamp during which an apelin infusion will be administered followed by a wash-out period and then, a second clamp in which a placebo infusion will be administered
  Interventions: Drug: apelin; Drug: placebo
- Placebo then Apelin (Other): First clamp during which a placebo infusion will be administered followed by a wash-out period and then, a second clamp in which an apelin infusion will be administered
  Interventions: Drug: apelin; Drug: placebo

INTERVENTIONS:
Drug: apelin — Assessing the difference between the insulin sensitivity measured during hyperinsulinemic euglycemic clamps in the presence of a 2 hours continuous infusion of (PYR1)-apelin-13 (30nmol/kg) versus a 2 hours continuous infusion of placebo (vehicle alone).
  Other Names: [pyr1]-apelin-13 infusion
Drug: placebo — 2 hours continuous infusion of placebo (vehicle alone) to compare with 2 hours infusion of apelin

SUMMARY:
Preclinical studies have demonstrated in mouse models that (PYR1)-apelin-13 exerts a glucose-regulating action in vivo. The (PYR1)-apelin-13 effect on insulin sensitivity in healthy overweighed volunteers has been previously assessed in a phase I clinical trial (APELINS study; NCT02033473). The APELINS-2 clinical trial aims to expand the initial proof of concept to the population targeted by future innovative insulin-sensitizing therapies: patients living with type 2 diabetes.

DETAILED DESCRIPTION:
Insulin sensitivity is measured using the hyperinsulinemic euglycemic glucose clamp method. The hypothesis of the investigators is that a continuous (pyr1)-apelin-13 infusion improves insulin sensitivity of type 2 diabetic patients compared to placebo infusion.

This study could bring new elements for understanding the pathophysiology of insulin resistance and type 2 diabetes mellitus in humans and could lead to the development of innovative therapies in type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type2 diabetes
* Body Mass Index between 27 and 33 kg / cm ²
* HbA1c < 8.5%
* Non-pathological Electrocardiogram
* Heart rate between 50 and 80 beats per minute at rest.
* Complete Blood Count (CBC) with no significant anomaly in terms of the investigator..
* Serum electrolytes without clinically significant abnormalities in terms of the investigator.
* Liver function tests without clinically significant abnormalities in terms of the investigator
* Renal function tests without clinically significant abnormalities in terms of the investigator
* Good peripheral vein (forearm and back of the hand).
* Agreement to participate in the establishment of a serum bank.
* Ability to sign informed consent.
* Affiliation to a social security scheme

Exclusion Criteria:

* Secondary prevention of cardio-vascular disease
* Insulin therapy or Glucagon Like Peptid 1 (GLP-1) analogs therapy in the 6 months before inclusion.
* Risk factor, treatment or electrocardiogram as recommended by International Conference on Harmonization (ICH) E14 "Clinical Evaluation of QT / QTc Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs"
* Repeated a QTc interval> 450 ms measurement
* Risk factor for torsade de pointes: myocardial infarction, hypokalemia, family history of long QT syndrome
* Personal history of cancer.
* Positive HIV serology.
* Hepatitis B serology positive.
* Positive hepatitis C serology.
* Cognitive impairment or mental illness (at the discretion of the investigator).
* Chronic excessive alcohol consumption (consumption > 30g/day or 210g/week).
* Person under judicial protection, guardianship.
* Subject with a resting systolic blood pressure greater than 140 mm Hg and diastolic blood pressure greater than 90 mmHg
* Smoking more than 10 cigaret per day and can not be interrupted for 24 hours.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Delta between Glucose Infusion Rate | 240 minutes
  Difference between glucose infusion rate measured during investigational product infusion (mean of values measured at 210, 215, 220, 225, 230, 235 and 240 minutes) and basal glucose infusion rate (mean of values measured at 90, 95, 100, 105, 110, 115 and 120 minutes).

SECONDARY OUTCOMES:
Measure of M-value (a glucose physiological parameter) | 240 minutes
  Difference between value of product time (mean of values measured at 210, 215, 220, 225, 230, 235 and 240 minutes) and value of basal (mean of values measured at 90, 95, 100, 105, 110, 115 and 120 minutes).
systolic blood pressure and diastolic blood pressure | 240 minutes
heart rate | 240 minutes
Measure of QTc interval with electrocardiogram examination | 240 minutes
Clinic sign of apelin intolerance | 240 minutes
Dosage of plasma proteins | 240 minutes
  A kinetic is realized with samples at 0, 15, 30, 45, 60, 75, 90, 100, 110, 120, 135, 150, 165, 180, 195, 200, 220, 230 and 240 minutes
Clinic sign of apelin allergy | 240 minutes
  Modification in physiological parameters
Clinic sign of apelin toxicity | 240 minutes
  Modification in physiological parameters

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Gourdy, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospitals of Toulouse (Rangueil), Toulouse, Midi-Pyrénées, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gourdy P, Cazals L, Thalamas C, Sommet A, Calvas F, Galitzky M, Vinel C, Dray C, Hanaire H, Castan-Laurell I, Valet P. Apelin administration improves insulin sensitivity in overweight men during hyperinsulinaemic-euglycaemic clamp. Diabetes Obes Metab. 2018 Jan;20(1):157-164. doi: 10.1111/dom.13055. Epub 2017 Aug 10. PMID 28681996